CLINICAL TRIAL: NCT00257257
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dose (Rimonabant 20 mg) Multicenter Study of Long-Term Glycemic Control With Rimonabant in Treatment-naïve Patients With Type 2 Diabetes
Brief Title: Study Evaluating Rimonabant Efficacy in Drug-NAive DiabEtic Patients
Acronym: SERENADE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5825
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Rimonabant (SR141716)

SUMMARY:
Primary: Effect on HbA1c over 6 months in drug-naive patients with type 2 diabetes

Secondary: Effect on glucose, insulin, C-peptide, insulin resistance, body weight, HDL-cholesterol, triglycerides, blood pressure - Safety, tolerability

DETAILED DESCRIPTION:
The total duration of the study will be up to 6 and 1/2 months including screening period (up to 14 days) and double-blind treatment period (approximately 6 months) in patients on mild hypocaloric diet (600 kcal/day deficit).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged greater than or equal to 18 years.
* Diagnosis of type 2 diabetes as defined by WHO criteria for at least 2 months but no longer than 3 years.
* Type 2 diabetes not previously treated by a pharmacological agent.

Note:

* a) insulin use is accepted if it is not within 6 months prior to screening visit and only for the following reasons:

  * prior use for management of gestational diabetes,
  * short-term (less than or equal to 1 month) use to maintain glycemic control for hospitalization, medical procedures, or intervention.
* b) use of an oral antidiabetic agent is accepted if it is not within 6 months prior to screening visit and only if it was prescribed for no more than 4 months.
* HbA1C greater than or equal to 7% and less than or equal to 10%.
* Having signed the informed consent form.

Exclusion Criteria:

General:

* Weight loss > 5 kg within 3 months prior to screening visit.
* Pregnancy or lactation.
* Absence of medically approved contraceptive methods for females of childbearing potential.
* Marijuana or hashish users.
* Administration of other investigational drugs within 30 days prior to screening visit.
* Previous participation in a rimonabant study.
* Presence or history of allergic reaction or intolerance to multiple drugs.
* Presence of any other condition (e.g., geographic, social) that the Investigator feels that would restrict or limit the patient's participation for the duration of the study.

Related to endocrine and metabolic disorders:

* Presence of any clinically significant endocrine disease according to the Investigator.

Note: euthyroid patients on replacement therapy will be included if the dosage of thyroxine is stable for at least 3 months prior to screening visit.

* Fasting C-peptide < 1.0 ng/mL.

Related to other disorders:

* Presence of any severe medical or psychological condition that in the opinion of the Investigator would compromise the patient's safety or successful participation in the study.
* Presence or history of cancer within the past five years with the exception of adequately treated localized basal cell skin cancer or in situ uterine cervical cancer.

Related to laboratory findings:

* Positive test for hepatitis B surface antigen and/or hepatitis C antibody.
* Abnormal TSH level (TSH > ULN or < LLN).
* Hemoglobin < 11 g/dL and/or neutrophils < 1,500/mm3 and/or platelets < 100,000/mm3.
* Positive urine pregnancy test.
* Positive urine test for marijuana or hashish metabolites.

Related to previous or concomitant medications:

* Oral antidiabetic agent except if it is not within 6 months prior to screening visit and only if it was prescribed for no more than 4 months.
* Insulin except if it is not within 6 months prior to screening visit and only for management of gestational diabetes or short-term use to maintain glycemic control for hospitalization, medical procedures, or intervention.
* Drugs affecting weight (e.g., sibutramine, orlistat, herbal preparations, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2005-03; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Absolute change in HbA1C from baseline to Month 6.

SECONDARY OUTCOMES:
Fasting glucose, fasting insulin, C-peptide, HOMA analysis, body weight, HDL-cholesterol, triglycerides, blood pressure, safety (physical examination, vital signs, laboratory tests, adverse events).

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Warsaw, Poland